CLINICAL TRIAL: NCT06155942
Title: Early Biomarkers of Neurodegeneration in Parkinsonian Syndromes: Analysis in Very High Field (7T) Brain MRI.
Brief Title: Early Biomarkers of Neurodegeneration in Parkinsonian Syndromes
Acronym: SODIPARK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RCAPHM22_0291; ID-RCB (Other: 2023-A01146-39)
Record Dates: First submitted 2023-11-17; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Parkinson Disease; Progressive Supranuclear Palsy
Keywords: MRI; Parkinson disease; progressive supranuclear palsy; biomarkers
MeSH Terms: conditions — Parkinson Disease; Supranuclear Palsy, Progressive | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with Parkinson Disease (Other)
  Interventions: Procedure: 7 Tesla MRI
- Patients with Progressive Supranuclear Palsy (Other)
  Interventions: Procedure: 7 Tesla MRI
- Healthy volunteers (Other)
  Interventions: Procedure: 7 Tesla MRI

INTERVENTIONS:
Procedure: 7 Tesla MRI — Patients will have a 7T MRI and questionnaires
  Other Names: Questionnaires

SUMMARY:
Parkinson's disease (PD) is the most common degenerative Parkinson's syndrome and is linked, among other things, to the excessive accumulation of an abnormally aggregating protein, alpha-synuclein. Progressive Supranuclear Palsy (PSP) is another Parkinson's syndrome, linked, among other things, to the abnormal accumulation of the protein Tau, and expressed clinically by falls, early cognitive impairment and oculomotor disorders, not present in PD. The onset of these disorders is so gradual that differential diagnosis between the two diseases is only possible at a late stage, on average 3 to 5 years after the onset of symptoms.

To date, there is a lack of validated imaging biomarkers for diagnosing and monitoring PD and PSP. There is therefore an urgent need for the development of robust biomarkers capable of detecting neurodegeneration at an early stage, in order to aid differential diagnosis as soon as symptoms appear, and to potentially enable these patients to be included in specific therapeutic trials (as these diseases are pathophysiologically different) with potential neuroprotective effects.

The development of cutting-edge technologies such as 7T MRI, combined with optimized image processing methods, now enable non-invasive in vivo exploration and analysis of these small structures in terms of ion homeostasis (sodium), microstructure (volumetry, amount of iron and neuromelanin) and connectivity.

ELIGIBILITY:
For Parkinson Disease:

Inclusion Criteria:

1. Patients aged between 40 and 80
2. Fulfilling the diagnostic criteria for MPI (Postuma et al., 2015)
3. First motor symptom (rigidity, akinesia, tremor) less than 36 months ago
4. Patient entitled to or affiliated with a social security scheme
5. Patients who understood, completed and signed the consent form for study participation.

Exclusion Criteria:

1. Patient with a neurological disease of the central nervous system other than those studied (including history of stroke, repeated head trauma, documented encephalitis). In case of doubt, this criterion will be left to the discretion of the principal investigator, who is a neurologist.
2. Contraindications to 7T MRI: presence of an ocular metallic foreign body (accidental shrapnel or other), pacemaker (cardiac simulator) or neurostimulator (pain treatment), cochlear implants or any implanted electronic medical equipment in general, metallic heart valve, vascular clips implanted on a cranial aneurysm.
3. Claustrophobia or any other condition preventing full MRI.
4. Montreal Cognitive Assessment (MOCA) test < 25/30
5. Pregnant or breast-feeding woman or protected person (under guardianship, curatorship, deprived of liberty).

For Progressive Supra-nuclear Palsy:

Inclusion criteria:

1. Patients aged 40 to 80
2. Fulfilling the diagnostic criteria for soPSP (Höglinger et al., 2017) :
3. First motor symptom (rigidity, akinesia, tremor) or falls or cognitive impairment (frontal syndrome or language disorder or cortico-basal syndrome) occurring less than 36 months ago
4. Patients benefiting from or affiliated to a social security scheme
5. Patients who have understood, completed and signed the study participation consent form

Exclusion criteria:

1. Patient with a neurological disease of the central nervous system other than those studied (including history of stroke, repeated head trauma, documented encephalitis). In case of doubt, this criterion will be left to the discretion of the principal investigator, who is a neurologist.
2. Contraindications to 7T MRI: presence of an ocular metallic foreign body (accidental shrapnel or other), pacemaker (cardiac simulator) or neurostimulator (pain treatment), cochlear implants or any implanted electronic medical equipment in general, metallic heart valve, vascular clips implanted on a cranial aneurysm.
3. Claustrophobia or any other condition preventing MRI.
4. Pregnant or breast-feeding woman or protected person (under guardianship, curatorship, deprived of liberty).

For Control group:

Inclusion criteria:

1. Subjects aged between 40 and 80
2. Subjects benefiting from or affiliated with a social security plan
3. Subjects who have understood, completed and signed the study participation consent form

Exclusion criteria:

1. Subjects with a known history of neurological disease of the central nervous system (e.g. Parkinson's disease, Alzheimer's, stroke, brain tumor, multiple sclerosis, amyotrophic lateral sclerosis, repeated head trauma, documented encephalitis, etc.). In case of doubt, this criterion will be left to the discretion of the principal investigator, who is a neurologist.
2. Contraindications to 7T MRI: presence of an ocular metallic foreign body (accidental shrapnel or other), pacemaker (cardiac simulator) or neurostimulator (pain treatment), cochlear implants or any implanted electronic medical equipment in general, metallic heart valve, vascular clips implanted on a cranial aneurysm.
3. Claustrophobia or any other condition preventing MRI.
4. Pregnant or breast-feeding women or protected persons (under guardianship, curatorship, deprived of liberty).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Sodium accumulation between Parkinson disease patients and Progressive Supranuclear Palsy | Between month 0 and month 3 after inclusion
  Comparison of intracerebral sodium accumulation measured by very high-field (7T) cerebral MRI between subjects with Idiopathic Parkinson's Disease and subjects with early-stage Progressive Supra-Nuclear Palsy

SECONDARY OUTCOMES:
Sodium accumulation between Parkinson disease patients (MPI) and control subjects | Between month 0 and month 3 after inclusion
  Comparison of intracerebral sodium accumulation between subjects with early-stage Parkinson's Disease (PD) and control subjects.
Sodium accumulation between Progressive Supra-nuclear patients (soPSP) and control subjects | Between month 0 and month 3 after inclusion
  Comparison of intracerebral sodium accumulation between subjects with soPSP and control subjects.
Brain atrophy between MPI and soPSP patients | Between month 0 and month 3 after inclusion
  3D mapping of brain atrophy differences measured in Voxel Based Morphometry (VBM), value in cm3
Brain atrophy between MPI and control group | Between month 0 and month 3 after inclusion
  3D mapping of brain atrophy differences measured in Voxel Based Morphometry (VBM), value in cm3
Brain atrophy between soPSP and control group | Between month 0 and month 3 after inclusion
  3D mapping of brain atrophy differences measured in Voxel Based Morphometry (VBM), value in cm3
Iron accumulation between soPSP and control group | Between month 0 and month 3 after inclusion
  3D mapping of iron accumulation differences measured by Quantitative Susceptibility Mapping (QSM), values in ppm
Iron accumulation between MPI and soPSP patients | Between month 0 and month 3 after inclusion
  3D mapping of iron accumulation differences measured by Quantitative Susceptibility Mapping (QSM), values in ppm
Iron accumulation between soPSP patients and control group | Between month 0 and month 3 after inclusion
  3D mapping of iron accumulation differences measured by Quantitative Susceptibility Mapping (QSM), values in ppm
Accumulation of neuromelanin between MPI and soPSP patients | Between month 0 and month 3 after inclusion
  3D mapping of neuromelanin differences (signal/MT ratio)
Accumulation of neuromelanin between MPI patients and control group | Between month 0 and month 3 after inclusion
  3D mapping of neuromelanin differences (signal/MT ratio)
Accumulation of neuromelanin between soPSP patients and control group | Between month 0 and month 3 after inclusion
  3D mapping of neuromelanin differences (signal/MT ratio)
Movement of water molecules between MPI and soPSP patients | Between month 0 and month 3 after inclusion
  3D mapping of differences in mean diffusivity (DM), values in mm2/s
Movement of water molecules between MPI patients and control group | Between month 0 and month 3 after inclusion
  3D mapping of differences in mean diffusivity (DM), values in mm2/s
Movement of water molecules between soPSP patients and control group | Between month 0 and month 3 after inclusion
  3D mapping of differences in mean diffusivity (DM), values in mm2/s
Structural connectivity between MPI and soPSP patients | Between month 0 and month 3 after inclusion
  3D mapping of anisotropy fraction (AF) differences, values between 0 and 1
Structural connectivity between soPSP patients and control group | Between month 0 and month 3 after inclusion
  3D mapping of anisotropy fraction (AF) differences, values between 0 and 1
Structural connectivity between MPI patients and control group | Between month 0 and month 3 after inclusion
  3D mapping of anisotropy fraction (AF) differences, values between 0 and 1
Measurement of the dependency between sodium accumulation and age | Between month 0 and month 3 after inclusion
  Correlation between sodium concentration (mmol/L) and age
Measurement of the dependency between sodium accumulation and sex | Between month 0 and month 3 after inclusion
  Correlation between sodium concentration (mmol/L) and sex
Measurement of the dependency between sodium accumulation and laterality | Between month 0 and month 3 after inclusion
  Correlation between sodium concentration (mmol/L) and laterality
Measurement of the dependency between brain atrophy and sex | Between month 0 and month 3 after inclusion
  Measure by Voxel Based Morphometry (VBM) in cm3 and sex
Measurement of the dependency between brain atrophy and age | Between month 0 and month 3 after inclusion
  Measure by Voxel Based Morphometry (VBM) in cm3 and age
Measurement of the dependency between brain atrophy and laterality | Between month 0 and month 3 after inclusion
  Measure by Voxel Based Morphometry (VBM) in cm3 and laterality
Measurement of the dependency between iron accumulation and age | Between month 0 and month 3 after inclusion
  Measure by Quantitative Susceptibility Mapping (QSM) in ppm and age
Measurement of the dependency between iron accumulation and sex | Between month 0 and month 3 after inclusion
  Measure by Quantitative Susceptibility Mapping (QSM) in ppm and sex
Measurement of the dependency between iron accumulation and laterality | Between month 0 and month 3 after inclusion
  Measure by Quantitative Susceptibility Mapping (QSM) in ppm and laterality
Measurement of the dependency between accumulation of neuromelanin and age | Between month 0 and month 3 after inclusion
  Correlation between ratio of signal/MT and age
Measurement of the dependency between accumulation of neuromelanin and sex | Between month 0 and month 3 after inclusion
  Correlation between ratio of signal/MT and sex
Measurement of the dependency between accumulation of neuromelanin and laterality | Between month 0 and month 3 after inclusion
  Correlation between ratio of signal/MT and laterality
Measurement of the dependency between structural connectivity and age | Between month 0 and month 3 after inclusion
  Correlation between anisotropy fraction (AF) and age
Measurement of the dependency between structural connectivity and sex | Between month 0 and month 3 after inclusion
  Correlation between anisotropy fraction (AF) and sex
Measurement of the dependency between structural connectivity and laterality | Between month 0 and month 3 after inclusion
  Correlation between anisotropy fraction (AF) and laterality
Measurement of the dependency between structural connectivity and duration of disease progression | Between month 0 and month 3 after inclusion
  Correlation between anisotropy fraction (AF) and duration of the disease
Measurement of the dependency between accumulation of neuromelanin and duration of disease progression | Between month 0 and month 3 after inclusion
  Correlation between ratio of signal/MT and duration of the disease
Measurement of the dependency between iron accumulation and duration of disease progression | Between month 0 and month 3 after inclusion
  Measure by Quantitative Susceptibility Mapping (QSM) in ppm and duration of the disease
Measurement of the dependency between brain atrophy and duration of disease progression | Between month 0 and month 3 after inclusion
  Measure by Voxel Based Morphometry (VBM) in cm3 and duration of disease progression
Measurement of the dependency between sodium accumulation and duration of disease progression | Between month 0 and month 3 after inclusion
  Correlation between sodium concentration (mmol/L) and duration of disease
Measurement of the dependency between sodium accumulation and sense of smell | Between month 0 and month 3 after inclusion
  Correlation between sodium concentration (mmol/L) and sense of smell (questionnaire)
Measurement of the dependency between brain atrophy and sense of smell | Between month 0 and month 3 after inclusion
  Measure by Voxel Based Morphometry (VBM) in cm3 and sense of smell (questionnaire)
Measurement of the dependency between iron accumulation and sense of smell | Between month 0 and month 3 after inclusion
  Measure by Quantitative Susceptibility Mapping (QSM) in ppm and sense of smell (questionnaire)
Measurement of the dependency between accumulation of neuromelanin and sense of smell | Between month 0 and month 3 after inclusion
  Correlation between ratio of signal/MT and sense of smell (questionnaire)
Measurement of the dependency between structural connectivity and sense of smell | Between month 0 and month 3 after inclusion
  Correlation between anisotropy fraction (AF) and sense of smell (questionnaire)
Measurement of the dependency between structural connectivity and severity of disease | Between month 0 and month 3 after inclusion
  Unified Parkinson's Disease Rating Scale (UPDRS), 0 to 199, 0 means better outcome
Measurement of the dependency between structural connectivity and quality of life | Between month 0 and month 3 after inclusion
  Schwab & England score, 0 to 100%, 0 means better outcome
Measurement of the dependency between accumulation of neuromelanin and quality of life | Between month 0 and month 3 after inclusion
  Schwab & England score, 0 to 100%, 0 means better outcome
Measurement of the dependency between iron accumulation and quality of life | Between month 0 and month 3 after inclusion
  Schwab & England score, 0 to 100%, 0 means better outcome
Measurement of the dependency between brain atrophy and quality of life | Between month 0 and month 3 after inclusion
  Schwab & England score, 0 to 100%, 0 means better outcome
Measurement of the dependency between sodium accumulation and quality of life | Between month 0 and month 3 after inclusion
  Correlation between Schwab & England score (Schwab & England score, 0 to 100%, 0 means better outcome) and sodium concentration (mmol/L)
Measurement of the dependency between accumulation of neuromelanin and severity of disease | Between month 0 and month 3 after inclusion
  Unified Parkinson's Disease Rating Scale (UPDRS), 0 to 199, 0 means better outcome
Measurement of the dependency between iron accumulation and severity of disease | Between month 0 and month 3 after inclusion
  Unified Parkinson's Disease Rating Scale (UPDRS), 0 to 199, 0 means better outcome
Measurement of the dependency between brain atrophy and severity of disease | Between month 0 and month 3 after inclusion
  Unified Parkinson's Disease Rating Scale (UPDRS), 0 to 199, 0 means better outcome
Measurement of the dependency between sodium accumulation and Hospital Anxiety and Depression | Between month 0 and month 3 after inclusion
  HAD Echelle (Hospital Anxiety and Depression), 0 to 3, 0 means better outcome
Measurement of the dependency between brain atrophy and Hospital Anxiety and Depression | Between month 0 and month 3 after inclusion
  HAD Echelle (Hospital Anxiety and Depression), 0 to 3, 0 means better outcome
Measurement of the dependency between iron accumulation and Hospital Anxiety and Depression | Between month 0 and month 3 after inclusion
  HAD Echelle (Hospital Anxiety and Depression), 0 to 3, 0 means better outcome
Measurement of the dependency between accumulation of neuromelanin and Hospital Anxiety and Depression | Between month 0 and month 3 after inclusion
  HAD Echelle (Hospital Anxiety and Depression), 0 to 3, 0 means better outcome
Measurement of the dependency between structural connectivity and Hospital Anxiety and Depression | Between month 0 and month 3 after inclusion
  HAD Echelle (Hospital Anxiety and Depression), 0 to 3, 0 means better outcome
Measurement of the dependency between structural connectivity and Sleep Behavior Disorder | Between month 0 and month 3 after inclusion
  REM Sleep Behavior Disorder Screening Questionnaire, 0 to 13, 0 means better outcome
Measurement of the dependency between accumulation of neuromelanin and Sleep Behavior Disorder | Between month 0 and month 3 after inclusion
  REM Sleep Behavior Disorder Screening Questionnaire, 0 to 13, 0 means better outcome
Measurement of the dependency between iron accumulation and Sleep Behavior Disorder | Between month 0 and month 3 after inclusion
  REM Sleep Behavior Disorder Screening Questionnaire, 0 to 13, 0 means better outcome
Measurement of the dependency between brain atrophy and Sleep Behavior Disorder | Between month 0 and month 3 after inclusion
  REM Sleep Behavior Disorder Screening Questionnaire, 0 to 13, 0 means better outcome
Measurement of the dependency between sodium accumulation and Sleep Behavior Disorder | Between month 0 and month 3 after inclusion
  REM Sleep Behavior Disorder Screening Questionnaire, 0 to 13, 0 means better outcome
Measurement of the dependency between sodium accumulation and motivation scale | Between month 0 and month 3 after inclusion
  Starkstein motivation scale, 0 to 42, 0 means worse outcome
Measurement of the dependency between brain atrophy and motivation scale | Between month 0 and month 3 after inclusion
  Starkstein motivation scale, 0 to 42, 0 means worse outcome
Measurement of the dependency between iron accumulation and motivation scale | Between month 0 and month 3 after inclusion
  Starkstein motivation scale, 0 to 42, 0 means worse outcome
Measurement of the dependency between accumulation of neuromelanin and motivation scale | Between month 0 and month 3 after inclusion
  Starkstein motivation scale, 0 to 42, 0 means worse outcome
Measurement of the dependency between structural connectivity and motivation scale | Between month 0 and month 3 after inclusion
  Starkstein motivation scale, 0 to 42, 0 means worse outcome
Measurement of the dependency between structural connectivity and non-motor fluctuations | Between month 0 and month 3 after inclusion
  Number of non-motor fluctuations
Measurement of the dependency between accumulation of neuromelanin and non-motor fluctuations | Between month 0 and month 3 after inclusion
  Number of non-motor fluctuations
Measurement of the dependency between iron accumulation and non-motor fluctuations | Between month 0 and month 3 after inclusion
  Number of non-motor fluctuations
Measurement of the dependency between brain atrophy and non-motor fluctuations | Between month 0 and month 3 after inclusion
  Number of non-motor fluctuations
Measurement of the dependency between sodium accumulation and non-motor fluctuations | Between month 0 and month 3 after inclusion
  Number of non-motor fluctuations
Measurement of the dependency between sodium accumulation and cognitives functions | Between month 0 and month 3 after inclusion
  Score Montreal Cognitive Assessment (MoCA), 0 to 30, 0 means worse outcome
Measurement of the dependency between brain atrophy and cognitives functions | Between month 0 and month 3 after inclusion
  Score Montreal Cognitive Assessment (MoCA), 0 to 30, 0 means worse outcome
Measurement of the dependency between iron accumulation and cognitives functions | Between month 0 and month 3 after inclusion
  Score Montreal Cognitive Assessment (MoCA), 0 to 30, 0 means worse outcome
Measurement of the dependency between accumulation of neuromelanin and cognitives functions | Between month 0 and month 3 after inclusion
  Score Montreal Cognitive Assessment (MoCA), 0 to 30, 0 means worse outcome
Measurement of the dependency between structural connectivity and cognitives functions | Between month 0 and month 3 after inclusion
  Score Montreal Cognitive Assessment (MoCA), 0 to 30, 0 means worse outcome
Measurement of the dependency between structural connectivity and quality of life | Between month 0 and month 3 after inclusion
  Parkinson's Disease Questionnaire (PDQ 39), 0 to 156, 0 means better outcome
Measurement of the dependency between accumulation of neuromelanin and quality of life | Between month 0 and month 3 after inclusion
  Parkinson's Disease Questionnaire (PDQ 39), 0 to 156, 0 means better outcome
Measurement of the dependency between iron accumulation and quality of life | Between month 0 and month 3 after inclusion
  Parkinson's Disease Questionnaire (PDQ 39), 0 to 156, 0 means better outcome
Measurement of the dependency between brain atrophy and quality of life | Between month 0 and month 3 after inclusion
  Parkinson's Disease Questionnaire (PDQ 39), 0 to 156, 0 means better outcome
Measurement of the dependency between sodium accumulation and quality of life | Between month 0 and month 3 after inclusion
  Parkinson's Disease Questionnaire (PDQ 39), 0 to 156, 0 means better outcome
Measurement of the dependency between sodium accumulation and hypotension | Between month 0 and month 3 after inclusion
  Blood pressure test for orthostatic hypotension
Measurement of the dependency between brain atrophy and hypotension | Between month 0 and month 3 after inclusion
  Blood pressure test for orthostatic hypotension
Measurement of the dependency between iron accumulation and hypotension | Between month 0 and month 3 after inclusion
  Blood pressure test for orthostatic hypotension
Measurement of the dependency between accumulation of neuromelanin and hypotension | Between month 0 and month 3 after inclusion
  Blood pressure test for orthostatic hypotension
Measurement of the dependency between structural connectivity and hypotension | Between month 0 and month 3 after inclusion
  Blood pressure test for orthostatic hypotension
Measurement of the dependency between structural connectivity and hallucinations | Between month 0 and month 3 after inclusion
  Miami Questionnaire, 0 to 70, 0 means better outcome
Measurement of the dependency between accumulation of neuromelanin and hallucinations | Between month 0 and month 3 after inclusion
  Miami Questionnaire, 0 to 70, 0 means better outcome
Measurement of the dependency between iron accumulation and hallucinations | Between month 0 and month 3 after inclusion
  Miami Questionnaire, 0 to 70, 0 means better outcome
Measurement of the dependency between brain atrophy and hallucinations | Between month 0 and month 3 after inclusion
  Miami Questionnaire, 0 to 70, 0 means better outcome
Measurement of the dependency between sodium accumulation and hallucinations | Between month 0 and month 3 after inclusion
  Miami Questionnaire, 0 to 70, 0 means better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Francois Cremieux, Study Director — AP-HM
Locations (6):
- France (6):
  - Ch Pays D'Aix, Aix-en-Provence
  - Hôpital Privé La Casamance - Service de Neurologie, Aubagne
  - Centre Hospitalier Avignon - Service de Neurologie, Avignon
  - CENTRE HOSPITALIER UNIVERSITAIRE NICE - Service de Neurologie, Nice
  - CENTRE HOSPITALIER NIMES - Service de Neurologie, Nîmes
  - CENTRE HOSPITALIER SAINTE MUSSE - Toulon, Toulon